CLINICAL TRIAL: NCT06579053
Title: An Open-label, Randomized, Single-dose, Two-period Crossover Design on Evaluating the Bioequivalence of Spironolactone Tablets 100mg (by SPH Sine Pharmaceutical Laboratories Co.,Ltd) and ALDACTONE® Tablets 100mg (by GD SEARLE LLC) in Healthy Adult Volunteers Under Fasting and Fed Conditions
Brief Title: Bioequivalence Study of Spironolactone Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SPH Sine Pharmaceutical Laboratories Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CRC-C2009
Record Dates: First submitted 2024-08-26; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Bioequivalence Study
MeSH Terms: interventions — Spironolactone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test product (Experimental): Spironolactone Tablets, 100 mg/tablet, to be orally administered.
  Interventions: Drug: Spironolactone Tablets (Test)
- Reference product (Active Comparator): ALDACTONE® Tablets,100 mg/tablet, to be orally administered.
  Interventions: Drug: Spironolactone Tablets (Reference)

INTERVENTIONS:
Drug: Spironolactone Tablets (Test) — Take one test tablet each period
  Arms: Test product
Drug: Spironolactone Tablets (Reference) — Take one reference tablet each period
  Other Names: ALDACTONE® tablets
  Arms: Reference product

SUMMARY:
The goal of this clinical trial is to Evaluate the Bioequivalence of Spironolactone Tablets 100mg (by SPH Sine Pharmaceutical Laboratories Co.,Ltd) and ALDACTONE® tablets 100mg (by GD SEARLE LLC) in Chinese Healthy Adult Volunteers under Fasting and Fed Conditions. It will also learn about the safety of the two drugs.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old ≤ age ≤ 40 years old, male or female;
2. Weight: ≥ 50 kg for male and ≥ 45 kg for female; body mass index (BMI) in the range of 19-26 kg/m2 (including 19 and 26);
3. No history of heart, liver, kidney, gastrointestinal, nervous system, mental abnormalities and metabolic abnormalities, no history of allergy to agents, no history of serious infections and serious injuries, etc;
4. Physical examination, vital signs examination, electrocardiogram examination, and laboratory examination of important indicators are normal or within the range considered acceptable by the sponsor/investigator;
5. No parenting plan and access to reliable contraception during the trial and within 3 months of the last dose;
6. Fully understand the purpose and requirements of the trial, voluntarily participate in the clinical trial and sign the ICF, and be able to complete the entire trial process according to the trial requirements.

Exclusion Criteria:

1. Persons with a known history of allergy, allergic disorder or hypersensitivity to the test product and any of its components or related agents;
2. Persons with a clear history of central nervous system, cardiovascular system, digestive system, respiratory system, urinary system, hematological system, metabolic disorders (e.g. hyperkalemia) or other diseases that are not suitable for participation in clinical trials (e.g. history of psychiatric disorders, etc.);
3. Those who have donated blood or lost ≥ 400 mL of blood within 3 months prior to enrollment;
4. Those who have taken any medication within 2 weeks prior to screening;
5. Those who have participated in other drug clinical trials within 3 months prior to enrollment;
6. current or former drug abuser or alcohol addict who consumes alcohol at least 2 times a day or 14 or more times a week, or is an avid drinker (1 drink defined as 125 mL of wine, 220 mL of beer or 50 mL of liquor; alcoholism defined as 5 or more drinks in approximately 2 hours);
7. Those who smoked more than 10 cigarettes per day during the 3 months prior to screening;
8. Hepatitis B surface antigen (HBsAg), HCV antibodies, syphilis spirochete antibodies and HIV antibody-positive persons;
9. Those with positive drug abuse screening results or alcohol breath test results;
10. Those with positive pregnancy test results(female)；
11. Those who have other factors that the investigator considers unsuitable for participation in the trial.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-08-23 (Actual)

PRIMARY OUTCOMES:
Cmax | up to 24 hours after tablet intake
  Maximum Observed Concentration in Plasma
AUC 0-t | up to 24 hours after tablet intake
  Area Under the Concentration-time Curve From Time Zero to Time of Last
AUC 0-∞ | up to 24 hours after tablet intake
  Area Under the Concentration-time Curve From Time Zero to Infinity

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No